CLINICAL TRIAL: NCT04224974
Title: Emotion and Symptom-Focused Engagement (EASE): A Multi-Site Randomized Controlled Trial of an Intervention for Individuals With Acute Leukemia
Brief Title: Emotion and Symptom-Focused Engagement Trial for Individuals With Acute Leukemia
Acronym: EASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Princess Margaret Hospital, University Health Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SC26
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Other: Usual Care (Experimental)
  Interventions: Other: Usual Care
- Behavioral: Usual Care + EASE Intervention-psy (Experimental): EASE Intervention = EASE-psy + EASE-phys
  Interventions: Behavioral: EASE-psy

INTERVENTIONS:
Other: Usual Care — The usual care group will receive usual care of their acute leukemia at their centre but no formal psychological or palliative care intervention as part of this trial
  Arms: Other: Usual Care
Behavioral: EASE-psy — All patients randomized to EASE will receive tailored supportive psychotherapy over the initial 8 weeks following the diagnosis of acute leukemia. The psychotherapy will be delivered by trained therapists and combines elements of relational support, affect regulation, and trauma-informed cognitive behavioural therapy (CBT).
  -EASE-phys: All patients randomized to EASE will receive weekly symptom screening during the initial inpatient treatment period (typically 4 weeks) with triggered referral to early palliative care (symptom control) to help manage moderate to severe physical symptoms based on a philosophy of multidisciplinary care and comprehensive assessment of symptoms.
  Arms: Behavioral: Usual Care + EASE Intervention-psy

SUMMARY:
The purpose of this study is to find out whether a novel manualized intervention, called Emotion and Symptom-focused Engagement (EASE), that combines psychological support with symptom screening plus triggered referral to early palliative care for symptom control, reduces psychological distress and physical symptom burden in individuals newly diagnosed with acute leukemia. To do this, half of the participants in this study will receive the usual care offered to patients with acute leukemia and half of the participants will receive usual care plus the EASE intervention.

DETAILED DESCRIPTION:
The standard or usual care treatment for patients with newly diagnosed acute leukemia involves admission to hospital for treatment (e.g. induction chemotherapy). Additional support services may be delivered if requested or if a doctor thinks it is necessary.

Little research has been done looking at the psychological and physical consequences of being diagnosed with and treated for acute leukemia, but our research team has found that a significant number of these individuals experience symptoms of traumatic stress and severe physical symptoms. Even less research has been done looking at ways to help alleviate this psychological and physical distress. Emotion and Symptom-focused Engagement (EASE) is an integrated psychosocial and early palliative care (symptom control) intervention designed to reduce psychological distress and physical symptom burden in patients newly diagnosed with acute leukemia. The EASE intervention provides i) tailored supportive psychotherapy (called EASE-psy) during the initial weeks of treatment to reduce symptoms of traumatic stress, and ii) symptom screening during the initial inpatient treatment period with triggered referral to early palliative care (symptom control) to help manage moderate to severe physical symptoms (called EASE-phys).

A phase II trial of EASE in patients with newly diagnosed acute leukemia demonstrated feasibility and preliminary evidence that it reduces psychological distress and physical symptom severity compared to usual care. This new trial is a definitive phase III, multi-site randomized controlled trial to test the effectiveness of EASE at reducing psychological distress and physical burden.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AL (acute myeloid leukemia (AML) and acute lymphocytic leukemia (ALL) chronic myelogenous leukemia (CML) in blast crisis; T-cell leukemia lymphoma (TLL), and AL of ambiguous lineage) and is recruited up to 1 week prior to hospital admission or within 2 weeks of hospital admission. For patients diagnosed with a mixed phenotype AL, the dominant sub-type must be identified for stratification purposes.
* Receiving or expected to receive induction therapy with curative intent at the time of recruitment.
* Age ≥ 18 years.
* Ability to pass the cognitive screening test at the time of recruitment (Short Orientation-Memory-Concentration Test (SOMC) score ≥ 20), unless deemed suitable at the CRA's discretion (e.g. in extenuating circumstances such as interruptions during the administration of the measure or when patients report a learning disability that can influence the results).
* Patient is fluent in English and is able (i.e. sufficiently literate and competent) and willing to complete the baseline questionnaires in English. Ability but unwillingness to complete the baseline questionnaires will make the patient ineligible.

Exclusion Criteria:

* Major communication difficulties at the time of recruitment, as assessed by the research team (e.g. severe hearing impairment or inability to speak).
* Receiving on-site (in hospital) psychological/psychiatric counseling at the time of recruitment.
* Receiving on-site (in hospital) palliative care services at the time of recruitment.
* A diagnosis of acute promyelocytic leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of the EASE intervention compared to usual care to reduce traumatic stress symptoms using the Stanford Acute Stress Reaction questionnaire (SASRQ) | 4 weeks
  This 30-item measure assesses severity of traumatic stress symptoms over the past four weeks; it has been updated to be Diagnostic and Statistical Manual of Mental Disorders (DSM-5)-concordant [American Psychiatric Association 2013] for acute stress disorder (ASD). Mean severity of traumatic stress symptoms at 4 weeks will be the first primary outcome
Assess the effect of the EASE intervention compared to usual care to reduce physical symptom severity using the Memorial Symptom Assessment Scale (MSAS) | 4 weeks
  This reliable and valid instrument assesses symptom prevalence, severity and distress associated with 26 common physical and 6 psychological symptoms of cancer. Mean physical symptom severity at 4 weeks will be the second primary outcome

SECONDARY OUTCOMES:
Assess the effect of the EASE intervention compared to usual care to reduce traumatic stress symptoms using the SASRQ | 8 weeks, 12 weeks & 26 weeks
Assess the effect of the EASE intervention to usual care to reduce physical symptom severity using the MSAS | 8 weeks, 12 weeks & 26 weeks
Assess the effect of the EASE intervention compared to usual care on the number of participants meeting criteria consistent with a diagnosis of ASD and threshold ASD based on DSM-5 criteria using the SASRQ | 4, 8, 12 and 26 weeks
Assess the effect of the EASE intervention compared to usual care on Quality of Life using The Functional Assessment of chronic Illness Therapy-Spiritual Well-being Scale | 4, 8, 12, 26 and 52 weeks
  Individual subscales of the FACIT-Sp provide scores for physical, social/family, emotional, functional spiritual well-being
Assess the effect of the EASE intervention compared to usual care on depressive symptoms using The Patient Health Questionnaire-9 (PHQ-9) | 4, 8 ,12 and 26 weeks
  This valid 9-item measure of depression has been widely used with patients with advanced cancer. Two additional items assessing intent to cause self-harm and interference with daily activities were included in the measure to ensure patients' safety but are not considered for data analysis.
Assess the effect of the EASE intervention compared to usual care on the number of physical symptoms of cancer and the associated symptom-related distress as measured by the (MSAS) | 4, 8, 12 & 26 weeks
Assess the effect of the EASE intervention compared to usual care on patient satisfaction with care using the 16-item FAMCAR-P16 | 4, 8, 12 and 26 weeks
Assess the effect of the EASE intervention compared to usual care on pain using the modified Brief Pain Inventory-Sort Form (BPI) | 4, 8 12 and 26 weeks
  The BPI is a widely used measure to rapidly assess the severity of pain and its impact on functioning and will be assessed as part of the secondary outcomes
The modified brief Experiences in Close Relationships Scale (ECR-M16) is an instrument to measure attachment security or the ability to rely on close others for support when distressed. | Baseline
  It provides subscale scores assessing attachment anxiety (i.e. fear of abandonment) and attachment avoidance (i.e. defensive independence). The ECR-M16 will only be administered at baseline in both arms of the study.
10) The EQ-5D-5L will be used to measure generic health status so that it can be used to compute quality-adjusted life years (QALY) in an economic evaluation that compares the benefit and cost of the EASE intervention | 4, 8, 12, 26 and 52 weeks
To compare progression-free survival between treatment arms | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rodin, Study Chair — Princess Margaret Hospital, University Health Network; Camilla Zimmerman, Study Chair — Princess Margaret Hospital, University Health Network
Locations (5):
- Canada (5):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Subject to CCTG policy
URL: https://www.ctg.queensu.ca/public/policies